CLINICAL TRIAL: NCT06311006
Title: Safety Registry of a Fecal Microbiota Transplant Cohort (COSMIC-FMT)
Brief Title: Safety Registry of a Fecal Microbiota Transplant Cohort
Acronym: COSMIC-FMT
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K170103J; 2019-A02579-48 (Other: ANSM)
Record Dates: First submitted 2024-02-28; First posted 2024-03-15 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Clostridium Difficile Infections
Keywords: Clostridium Difficile Infection; Fecal microbiota transplantation
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma and stools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: adult patients for whom FMT for CDI is indicated and planned as part of the routine care (definition of CDI and recurrence according to European recommendations 2014 10)
- Stool donor

SUMMARY:
Clostridium difficile infection (CDI) is a major cause of infectious diarrhea and the most important cause of nosocomial diarrhea. Recurrent forms are a major problem with this infection. The use of fecal microbiota transplantation (FMT), FMT appears in the most recent European and North American recommendations.

There is no cohort or multicenter registry in France prospectively collecting FMTs, the methods used, their efficacy and side effects. Likewise, there is no prospective collection focused on the cohort of stool donors. A large national cohort of patients who have undergone FMT as part of routine care as well as donors, is essential for evaluating the safety of FMT.

DETAILED DESCRIPTION:
Clostridium difficile infection (CDI) is a major cause of infectious diarrhea and the most important cause of nosocomial diarrhea. For 20 years, the incidence of CDI has continued to increase. In addition, the severity of infections is also increasing (mortality: 5% in 1990 against 13.8% in 2003; complications: 6% in 1990 against 18% in 2003).

Recurrent forms represent a major problem of this infection. Indeed, after a first episode, the risk of a first recurrence is around 15 to 25% and this risk then increases with each recurrence, reaching 45% then 65% after a first and second recurrence respectively. These Recurrent forms pose a real therapeutic problem, causing significant morbidity (repeated hospitalizations, time off work, etc.) and substantial mortality. Patients with CDI are 2.5 times more likely to die within 30 days of infection than uninfected patients, regardless of age or comorbidities. The mortality rate is also higher in patients with a recurrent form than in those with a single episode. Furthermore, the antibiotics usually used are only marginally effective in cases of recurrent CDI.

Numerous studies, including two randomized trials, have shown that fecal microbiota transplantation (FMT), is superior to antibiotic therapy in reducing subsequent recurrences, the use of FMT in this indication appears in the most recent European and North American recommendations.

Cosmic-FMT cohort aims to be as representative as possible of the population of patients having FMT for CDI in the context of care.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* Adult patient with an indication for FMT for CDI (severe refractory CDI, recurrent CDI);
* Informed written consent

Donors:

* Adult (18 years or older)
* Informed Written consent

Exclusion Criteria:

* insufficient level of understanding of written and spoken French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with an indication for fecal microbiota transplantation as part of the treatment for Clostridium difficile infection
Sampling Method: Non-Probability Sample
Enrollment: 305 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2029-01-04 (Estimated); Study Completion 2029-01-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of hospitalizations attributable to FMT | Week 10 and 3 years after FMT

SECONDARY OUTCOMES:
Proportion of Clostridium difficile relapses | 10 weeks after FMT, and 3 years
  In the short term: rate of occurrence of at least one recurrence of CDI within 10 weeks after FMT; In the medium term: rate of occurrence of at least one recurrence of CDI > 10 weeks and ≤ 3 years after FMT.
Proportion of relapse | Week 10 and 3 years
  The strains will be characterized in each center according to local methods.
Proportion of reinfections | Week 10 and 3 years
  The strains will be characterized in each center according to local methods.
Efficacy of FMT in CDI (defined as free from relapse) at 10 weeks and 3 years according to clinical characteristics of donors | at 10 weeks and 3 years
Efficacy of FMT in CDI (defined as free from relapse) at 10 weeks and 3 years according to clinical characteristics of patients | at 10 weeks and 3 years
Efficacy of FMT in CDI (defined as free from relapse) at 10 weeks and 3 years according to the method of preparation and administration of fecal preparation | at 10 weeks and 3 years
Evolution of transit (i.e. number of stools per day and their consistency) and mean BMI in patients Correlation between the evolution of transit and the BMI of the donor and the patient. | Before and after FMT at Week 10, at Month 6 then every 6 months until Month 36
Patient status (absence of recurrence or relapse or re-infection) according to the composition of the microbiota (by sequencing or metabolomic method or culture) of the donors. | Week 10
Composition of the patient's microbiota before FMT and at week 10 and composition of the donor's microbiota (by sequencing or metabolomic method or culture) of the raw stool and the preparation to be administered to the patient. | before FMT and at week 10 for patients
adverse event rate | 24hours, 10weeks, every 6 months until 3 years
  In the short term, all adverse events occurring within 24 hours following FMT and within 10 weeks following FMT will be recorded based on both a predetermined list of events of interest as well as on an open declaration.
  In the medium term, potential adverse events in the patient will be recorded every 6 months for 3 years also based on a predetermined list of events and on an open declaration.
  Occurrence of at least one SAE at W10 and 3 years according to (i) the clinical characteristics of the donors, (ii) the clinical characteristics of the patients, (iii) the method of preparation and administration of the fecal preparation.
Metabolomic, immunological analysis (phenotype of peripheral blood immune cells) of the donor and the patient before and after FMT (at W10). | Day 0 and Week 10

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Department of Saint Antoine Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided